CLINICAL TRIAL: NCT02250482
Title: An Open Study to Investigate the Safety and Efficacy of Optivate® in Haemophilia A Patients Undergoing Surgery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 8VWF02
Record Dates: First submitted 2014-09-02; First posted 2014-09-26 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — optivate; Factor VIII

ARMS (1):
- Optivate® (Experimental): Optivate® (Human Coagulation Factor VIII)
  Interventions: Biological: Optivate® (Human Coagulation Factor VIII)

INTERVENTIONS:
Biological: Optivate® (Human Coagulation Factor VIII)

SUMMARY:
The main objective of the study is to investigate the safety and efficacy of Optivate®, administered in appropriate dosage to present bleeding and achieve haemostasis in patients with Haemophilia A undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Haemophilia A, at least 12 years of age, due to undergo surgery and have a lifetime exposure of at least 20 exposures to a FVIII concentrate.

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-11; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Incremental Recovery for plasma Factor VIII | 90 minutes after pre-operative bolus dose
  Incremental recovery is defined as peak rise in plasma Factor VIII levels divided by Factor VIII dose in IU/KG

CONTACTS AND LOCATIONS:
Locations (8):
- Poland (3):
  - Klinika Haematologii, Akademia Medyczna w Gdansku, ul., Debinki 7, 80-211 Gdansk
  - Klinika Haematologii, Akademia Medyczna w Lublinie, ul., Dr K Jaczewskiego 8, 20-090, Lublin
  - Klinika Haematologii, Akademia Medyczna w Poznaniu, ul., Szkolna 8/12, 61-833 Poznan
- United Kingdom (5):
  - Haemophilia Centre, Addenbrooke's Hospital, Hills Road, Cambridge
  - Haemophilia Centre, University Dept. of Haemophilia, Manchester Royal Infirmary, Manchester
  - Haemophilia Centre, University Hospital, Queens Medical Centre, Clifton Boulevard, Nottingham
  - Sheffield Haemophilia & Thrombosis Centre, Royal Hallamshire Hospital, Glossop Road, Sheffield
  - Haemophilia Centre, Southampton General Hospital, Tremona Road, Southampton

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk